CLINICAL TRIAL: NCT02763436
Title: "Improves Physiological Based Cord Clamping (PBCC) the Systemic and Cerebral Oxygenation in Term Infants?"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Schwaberger Bernhard, MD PhD, Ass.Dr. (MD) Mirjam Pocivalnik, Medical University of Graz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 28-078 ex 15/16
Record Dates: First submitted 2016-04-02; First posted 2016-05-05 (Estimated); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Near-Infrared Spectroscopy; Umbilical Cord Issue
Keywords: Neonatal transition; Umbilical cord clamping; Regional cerebral oxygen saturation; Cerebral blood volume; Near-infrared spectroscopy; Arterial oxygen saturation; Term infants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group "immediate cord clamping" (ICC) (No Intervention): The cord will be clamped within the first minute after birth, afterwards the newborn will be placed on the mothers chest/abdomen. This corresponds to the present routine approach in Graz.
- Group "physiological based cord clamping" (PBCC) (Active Comparator): The newborn will be placed on mother's chest/abdomen with intact cord. After the newborn has established stable breathing efforts (continuous regular breathing pattern and SpO2 values >25th percentile from Dawson et al "reference range for oxygen saturation" -minute 2>58%, minute 3>67%, minute 4>76%) the cord is clamped. This will need 2 - 4 minutes.
  Interventions: Procedure: physiological-based cord clamping

INTERVENTIONS:
Procedure: physiological-based cord clamping — The cord of the newborn infant is clamped after establishing stable breathing efforts. The suspected time ranges from 2-4 minutes.
  Arms: Group "physiological based cord clamping" (PBCC)

SUMMARY:
The first major intervention a newborn infant is facing following birth is clamping of the umbilical cord. This means separation of the infant from the placenta, the newborn becomes an independent individual, especially from a cardio-circulatory perspective. There is still a lack of understanding of the issues associated with umbilical cord clamping. The aim of the present study is to investigate whether cord clamping after onset of sufficient spontenous breathing is able to improve systemic and cerebral oxygenation in term infants delivered vaginally.

DETAILED DESCRIPTION:
Recent literature focused very much on the appropriate timing of the cord clamping (CC), distinguishing immediate cord clamping (ICC) from delayed cord clamping (DCC). Although potential benefits for DCC have been documented, especially for preterm infants, ICC still is the most widely used procedure. Although the reasons for this are unclear, a lack of understanding of the issues associated with umbilical cord clamping is thought to be a major underlying factor.

In animal research with fetal lambs it has been shown, that aeration of the lung played a crucial role in undisturbed cardio-circulatory immediate neonatal transition. Thus a new concept of DCC was introduced, delaying cord clamping until ventilation/aeration of the lung was established, calling this "Physiological-Based Cord Clamping" (PBCC). It was shown, that PBCC improved not only cardiovascular function in preterm lambs, but systemic and cerebral oxygenation too. Systemic oxygenation was measured using pulseoximetry, and cerebral oxygenation was measured using near infrared spectroscopy (NIRS).

Until now, human data for PBCC are lacking. Therefore, the aim of the present study is to investigate whether PBCC is able to improve systemic and cerebral oxygenation in term infants delivered vaginally.

ELIGIBILITY:
Inclusion Criteria:

* Vaginally born and term infants
* undisturbed transition period

Exclusion Criteria:

* congenital malformations
* respiratory support during transition period

Ages: 0 Minutes to 30 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2016-09-08 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Change in cerebral regional oxygen saturation (crSO2) | 15 minutes
  Difference in the course of postnatal increase of crSO2 (%). crSO2 is measured with nearinfrared spectroscopy (NIRS). Immediately after delivery, the NIRS sensor is placed on the left forehead, measuring crSO2 non-invasively over the observational period.

SECONDARY OUTCOMES:
Change in peripheral arterial oxygen saturation (SpO2) | 15 minutes
  Difference in the course of postnatal increase of SpO2 (%). SpO2 is measured with pulsoximetry, noninvasively. Immediately after delivery, the SpO2 sensor is placed on the right forearm/wrist to monitor peripheral preductal oxygen saturation over the observational period.
Change in Cerebral blood volume (CBV) | 15 minutes
  Differences in course of CBV decrease during the observational period. CBV (ml/100gbrain) is calculated out of data measured with NIRS noninvasively : depending on the changes of oxygenated and deoxygenated Hemoglobin.
Evaluation of cardiac shunt parameters | 20 minutes
  Collection of the following parameters using echocardiography: shuntdirection and diameter of the Ductus arteriosus and Foramen ovale.
Evaluation of preload parameters | 20 minutes
  Collection of the following parameters using echocardiography: superior vena cava (SVC) Flow and inferior vena cava (IVC) size.
right atrial (RA) and right ventricular (RV) dimension parameters | 20 minutes
  Collection of the following parameters using echocardiography: end-systolic right atrial size and area, end-diastolic plus end-systolic right ventricle size and area.
right ventricular (RV) systolic function | 20 minutes
  Calculation of the following parameters using echocardiography: TAPSE (tricuspid annular plane systolic excursion) as a measure of systolic right ventricular function.

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Schwaberger, MD PhD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhatt S, Polglase GR, Wallace EM, Te Pas AB, Hooper SB. Ventilation before Umbilical Cord Clamping Improves the Physiological Transition at Birth. Front Pediatr. 2014 Oct 20;2:113. doi: 10.3389/fped.2014.00113. eCollection 2014. PMID 25368858
- [Background] Bhatt S, Alison BJ, Wallace EM, Crossley KJ, Gill AW, Kluckow M, te Pas AB, Morley CJ, Polglase GR, Hooper SB. Delaying cord clamping until ventilation onset improves cardiovascular function at birth in preterm lambs. J Physiol. 2013 Apr 15;591(8):2113-26. doi: 10.1113/jphysiol.2012.250084. Epub 2013 Feb 11. PMID 23401615
- [Background] Hooper SB, Polglase GR, te Pas AB. A physiological approach to the timing of umbilical cord clamping at birth. Arch Dis Child Fetal Neonatal Ed. 2015 Jul;100(4):F355-60. doi: 10.1136/archdischild-2013-305703. Epub 2014 Dec 24. PMID 25540147
- [Background] Polglase GR, Dawson JA, Kluckow M, Gill AW, Davis PG, Te Pas AB, Crossley KJ, McDougall A, Wallace EM, Hooper SB. Ventilation onset prior to umbilical cord clamping (physiological-based cord clamping) improves systemic and cerebral oxygenation in preterm lambs. PLoS One. 2015 Feb 17;10(2):e0117504. doi: 10.1371/journal.pone.0117504. eCollection 2015. PMID 25689406
- [Background] Hooper SB, Harding R. Fetal lung liquid: a major determinant of the growth and functional development of the fetal lung. Clin Exp Pharmacol Physiol. 1995 Apr;22(4):235-47. doi: 10.1111/j.1440-1681.1995.tb01988.x. PMID 7671435
- [Background] Dawson JA, Kamlin CO, Vento M, Wong C, Cole TJ, Donath SM, Davis PG, Morley CJ. Defining the reference range for oxygen saturation for infants after birth. Pediatrics. 2010 Jun;125(6):e1340-7. doi: 10.1542/peds.2009-1510. Epub 2010 May 3. PMID 20439604
- [Derived] Schwaberger B, Ribitsch M, Pichler G, Krainer M, Avian A, Baik-Schneditz N, Ziehenberger E, Mileder LP, Martensen J, Mattersberger C, Wolfsberger CH, Urlesberger B. Does physiological-based cord clamping improve cerebral tissue oxygenation and perfusion in healthy term neonates? - A randomized controlled trial. Front Pediatr. 2023 Jan 9;10:1005947. doi: 10.3389/fped.2022.1005947. eCollection 2022. PMID 36699304